CLINICAL TRIAL: NCT02794740
Title: Study of X0002 Following Escalating Single and Multiple Doses Administered as Topical Application in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin XinChen-Techfields Pharma Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TFR-X0002-101
Record Dates: First submitted 2016-06-01; First posted 2016-06-09 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- X0002 First Dose (Experimental): Preliminary Experiment,4 Subjects,Single-Dose,Once,Non-Blind.
  Interventions: Drug: X0002
- X0002 Second Dose (Experimental): 8 Subjects,Single Dose once and Multiple Doses 7 Days,b.i.d,12 Hours Apart,Double-Blind.
  Interventions: Drug: X0002
- Placebo Second Dose (Placebo Comparator): 2 Subjects,Single Dose once and Multiple Doses 7 Days,b.i.d,12 Hours Apart,Double-Blind.
  Interventions: Drug: Placebo
- X0002 Third Dose (Experimental): 8 Subjects,Single Dose once and Multiple Doses 7 Days,b.i.d,12 Hours Apart,Double-Blind.
  Interventions: Drug: X0002
- Placebo Third Dose (Placebo Comparator): 2 Subjects,Single Dose once and Multiple Doses 7 Days,b.i.d,12 Hours Apart,Double-Blind.
  Interventions: Drug: Placebo
- X0002 Fourth Dose (Experimental): 8 Subjects,Single Dose,Once,Double-Blind.
  Interventions: Drug: X0002
- Placebo Fourth Dose (Placebo Comparator): 2 Subjects,Single Dose,Once,Double-Blind.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: X0002 — External Spray
  Arms: X0002 First Dose; X0002 Fourth Dose; X0002 Second Dose; X0002 Third Dose
Drug: Placebo — External Spray
  Arms: Placebo Fourth Dose; Placebo Second Dose; Placebo Third Dose

SUMMARY:
Primary Objectives:

To evaluate the safety and tolerability of escalating single and multiple doses of X0002 administered as a topical application.

Secondary Objectives:

To characterize the single and and multiple pharmacokinetics of escalating doses of X0002 and its active metabolite ibuprofen as a topical application.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male or female, each sex ratio does no less 1/3;
* Were between the ages of 18 and 45 years, inclusive. General condition is will;
* Were between the Body Mass Index (BMI) of 19-28, inclusive; BMI=Weight(kg)/Height2 (m2); Weight≥50kg (female) and 60kg (male);
* Nearly half of the year, no child care program and agree to take effective measures to contraception during the study period, blood pregnancy test of women in childbearing age was negative;
* Vital signs (measurement seated after resting 5 minutes) in the following range

  1. Temperature (auxiliary temperature): 35.0-37.0℃
  2. Systolic Pressure: 90-139mmHg
  3. Diastolic Pressure: 60-89mmHg
  4. sphygmus: 55-99bpm
* Subjects to fully understand the purpose, properties, method and reactions may occur of test drug trials. Were capable of giving informed consents voluntarily, and agreed to comply with the requirements of clinical protocols.

Exclusion Criteria:

* Primary disease in important organs;
* Mental or physical disability;
* Familial hereditary diseases;
* Clinically significant history of Electrocardiograph (ECG) abnormality, or Electrocardiograph (ECG) abnormality in the Screening or Baseline;
* Clinically significant abnormities in laboratory examination:

  1. Clinically significant abnormities in Liver Function Tests, for example aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) or bilirubin.
  2. Creatinine and Urea Nitrogen exceeded the upper limit of normal, or significant abnormities in urinary composition.
  3. Clinically significant abnormities of routine blood test, for example anemia, Leukocyte reduced, Platelet significantly reduced,etc.( Combined with adverse events in the laboratory to determine the value of abnormal).
  4. Abnormality of immunology, including HIV(human immunodeficiency virus) antibody positive, Hepatitis B surface antigen (HBsAg) positive, HCV(hepatitis C virus) antibody positive or Syphilis antibody positive.
* Drug abusers,or drug screening positive;
* Who was addicted to alcohol and tobacco (drinking 14 units of alcohol per week: 1 unit = beer 285 ml, or liquor 25 ml, or wine 1 cup. numbers of daily smoking ≥ 5) and / or not smoking and drinking in the test period;Test positive for nicotine or breath test positive for alcohol(>0.0mg/100ml);
* Took any drug long excretory phase that may affect the study, or in the past 3 months participated in any drug clinical trials;
* Entering the group 4 weeks ago used any prescription drugs ,or used any over the counter (OTC) drugs within 2 weeks (vitamins, herbal tonics, etc.), or before entering the group within 2 weeks took excessively food that effected drug metabolizing enzymes, such as grapefruit or grapefruit drink. Can the use of acetaminophen, but must record report in case report form (CRF）;
* A history of gastrointestinal bleeding or peptic ulcers, drugs allergy for aspirin or hypersensitivity to aspirin or other NSAIDs (Non-Steroidal Antiinflammatory Drugs), or a history of asthma or other allergic-type reactions after taking aspirin or other NSAIDs(Non-Steroidal Antiinflammatory Drugs); A history of intolerance or hypersensitivity to ibuprofenamine hydrochloride or any excipients or to the diluent ethanol;
* Donation or blood collection, or acute loss of blood during the 3 months prior to screening( more than 400ml);
* Had skin diseases wound or other symptom, investigators consider that maybe unsafe for subjects or effect of evaluation for application sites;
* There was a clinical significance history of allergy for drugs or food, or atopic allergic diseases (asthma, urticaria, eczema dermatitis) or a known drug allergy for test drugs or similar drugs;
* Lactating women, pregnant women or unable to take effective contraceptive measures;
* Researchers believed that participants not suitable to take the test for other factors.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Single Dose Arms:6days;Multiple Doses Arms:17days
  Adverse Event; Vital Signs; Physical Examination; Laboratory Examination; Electrocardiograph; Skin Irritation

SECONDARY OUTCOMES:
Pharmacokinetic parameters(Maximum Plasma Concentration [Cmax]) | Single Dose Arms:0-120hours;Multiple Doses Arms:0-120hours post-dose;11th day pre-dose;12th day 0-120 hours post-dose.

OTHER OUTCOMES:
Pharmacokinetic parameters(Area Under Curve [AUC]) | Single Dose Arms:0-120hours;Multiple Doses Arms:0-120hours post-dose;11th day pre-dose;12th day 0-120 hours post-dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Xinchen-Techfields Pharma Co. Ltd, Tianjin, Tianjin Municipality, China